CLINICAL TRIAL: NCT06229184
Title: Can Fecal Calprotectin Be Used as a Biomarker of Non-alcoholic Fatty Liver Disease In Obese Adolescents?
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sisli Hamidiye Etfal Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Busra Tetik Dincer, Resident doctor, Sisli Hamidiye Etfal Training and Research Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: 15.11.2022-2124
Record Dates: First submitted 2024-01-09; First posted 2024-01-29 (Actual); Last update posted 2024-02-13 (Actual); Status verified 2024-02

CONDITIONS: Obesity, Childhood; NAFLD
MeSH Terms: conditions — Pediatric Obesity; Non-alcoholic Fatty Liver Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control group (Experimental): Fecal calprotectin samples taken for comparison from healthy adolescents
  Interventions: Diagnostic Test: Fecal Calprotectin Test
- Obese group (Experimental): Fecal calprotectin samples taken from obese adolescents
  Interventions: Diagnostic Test: Fecal Calprotectin Test
- Obese + NAFLD group (Experimental): Fecal calprotectin samples taken from obese adolescents that have NAFLD
  Interventions: Diagnostic Test: Fecal Calprotectin Test

INTERVENTIONS:
Diagnostic Test: Fecal Calprotectin Test — Fecal samples are taken fom obese and healthy adolescents for study

SUMMARY:
The incidence of non-alcoholic fatty liver disease (NAFLD) is increasing with obesity, and it is believed that ongoing inflammation in obesity and alterations in the enterohepatic axis contribute to this process. This study aimed to determine the role of fecal calprotectin (FCP) as an inflammatory biomarker in course of obesity and NAFLD.

DETAILED DESCRIPTION:
Obesity is a significant public health issue worldwide. With the increasing prevalence of obesity, the prevalence of metabolic syndrome in adolescents is also on the rise. Non-alcoholic fatty liver disease (NAFLD), a major cause of chronic liver disease, is the hepatic component of metabolic syndrome. The prevalence of NAFLD is not precisely known, but in some studies, it is between 22.5% and 52.8% in children with obesity, constituting 2.6% of all children. Although the mechanisms involved in the development of obesity-related metabolic complications and NAFLD are not well understood, it is believed that intestinal inflammation, changes in the microbiota, and alterations in the gut-liver axis (GLA) may play a role in the development of low-grade chronic inflammation in NAFLD associated with obesity. Fecal calprotectin (FCP), which has become increasingly important in demonstrating intestinal inflammation in recent years, is a widely used test, particularly in the diagnosis and monitoring of inflammatory bowel disease and various gastrointestinal disorders. In our study, the utility of FCP as an inflammatory biomarker in the course of NAFLD in obese adolescents has been investigated. The study was approved by our hospital's ethics committee in 15.11.2022 and another ethics committee approval was taken in 08.06.2023 for title change of study. This study conducted under the Helsinki Declaration.

ELIGIBILITY:
Inclusion Criteria:

* 10-18 years old healthy adolescents for control group
* Children aged 10-18 years without any additional diseases, BMI>2 SD, no hepatosteatosis detected by ultrasonography (USG), and alanine aminotransferase (ALT) levels within normal limits were included in the obese group
* Children aged 10-18 years without any additional diseases, BMI>2 SD, Hepatosteatosis detected by ultrasonography (USG), and alanine aminotransferase (ALT) levels higher than normal limits adjusted for gender were included in the obese + NAFLD group

Exclusion Criteria:

* Diseases other than obesity and NAFLD

Ages: 10 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 41 (Actual)
Dates: Start 2022-11-16 (Actual); Primary Completion 2023-08-10 (Actual); Study Completion 2023-08-10 (Actual)

PRIMARY OUTCOMES:
Fecal Calprotectin Levels | Through study completion, an average of 3 months
  Fecal calprotectin levels expected to be higher in obese adolescents, even higher in obese + NAFLD adolescents

SECONDARY OUTCOMES:
Alanine Aminotransferase (ALT) Levels | Through study completion, an average of 3 months
  ALT levels expected to be higher in NAFLD adolescents

CONTACTS AND LOCATIONS:
Overall Officials: Ayşe Merve Usta, M.D., Study Director — Sisli Hamidiye Etfal Training and Research Hospital
Locations (1):
- Sisli Hamidiye Etfal Training and Research Hospital, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Dincer BT, Usta AM, Kural A, Helvaci N, Ucar A, Urganci N. Can fecal calprotectin be used as a biomarker of non-alcoholic fatty liver disease in obese adolescents? BMC Pediatr. 2024 Dec 23;24(1):834. doi: 10.1186/s12887-024-05327-4. PMID 39716084